CLINICAL TRIAL: NCT05048628
Title: The Effect of Ice, Green Tea and Arnica Montana Application on Post-Operative Intubation Related Sore Throat and Hoarseness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülcan Dürüst Sakallı, lecturer, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EasternMU-SBF-HB-GDS-01
Record Dates: First submitted 2021-07-13; First posted 2021-09-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2022-10

CONDITIONS: Sore Throat; Hoarseness
Keywords: green tea; arnico montana; ice Application; Endotracheal Intubation; Sore Throat; Nursing; Hoarseness
MeSH Terms: conditions — Pharyngitis; Hoarseness

STUDY DESIGN:
Intervention Model Description: Four Groups. Group were comprised of control group, green tea Gargle Solution group, ice pieces impregnated group, arnica montana tea Gargle Solution group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Multiple blinding (data collectors, participants, statistician, and reporters) was performed in the Randomized Controlled Experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- İce Pieces İmpregnated Group (Active Comparator): Impregnation of pieces of ice was delivered to us; one ice cube is planned after wearing and movements automatically by the throat purchase to exit use and sound program, and move with one ice cube after movement. It can be used after extubation. It is in sound class with Visual Analogue Scale (VAS) for the use of customers before and after the application. Extubation is in the last 0. hours, no small application is made, only in sound class with VAS. Evaluated by Stout's Hoarseness Scale
- Green Tea Gargle Solution Group (Active Comparator): To the patients included in the gargle group with green tea; four after, six after eigth after hours after extubation, the patients of the intervention group were asked to gargle 30 cc of green tea and before the application and after the patient's oral intake was requested by the physician to prevent sore throat and hoarseness afterwards, patients' sore throat is measured with Visual Analogue Scale (VAS) and hoarseness is measured with Stout's Hoarseness Scale. At the 0. th hour after extubation, no treatment is applied to the patients, only sore throat is evaluated with VAS and hoarseness is evaluated with Stout's Hoarseness Scale.0
- Arnica Montana Tea Gargle Solution Group (Active Comparator): To the patients included in the gargle group with arnica montana tea; four after, six after eigth after hours after extubation, the patients of the intervention group were asked to gargle 30 cc of arnica montana tea and before the application and after the patient's oral intake was requested by the physician to prevent sore throat and hoarseness afterwards, patients' sore throat is measured with Visual Analogue Scale (VAS) and hoarseness is measured with Stout's Hoarseness Scale. At the 0th hour after extubation, no treatment is applied to the patients, only sore throat is evaluated with VAS and hoarseness is evaluated with Stout's Hoarseness Scale.
- Control Group (No Intervention): Patients in the control group; sore throat and hoarseness scores at 0 hour immediately after extubation,to collect at 4, 6 and 8 hours after extubation, sore throat (Visual Analogue Scale) VAS; Stout s Voice if hoarseness It is evaluated with the Slightness Scale.

INTERVENTIONS:
Other: Comparıson — Only evaluation will be made at 0, 4, 6, and 8 hours after surgery without intervention in the control group.
  For other groups; Evaluation will be made at the 0th hour after the operation without application. The application will be made at the 4th, 6th, and 8th hours after the surgery and the resulting pain and hoarseness will be evaluated.

SUMMARY:
The study was planned to determine the effect of arnica montana, green tea mouthwash and ice particles impregnation on postoperative sore throat and hoarseness.

DETAILED DESCRIPTION:
Research Hypotheses Hl: Gargling with green tea after surgery reduces sore throat. H2: Impregnation of postoperative ice particles reduces sore throat. H3: Post-operative gargling with arnico montana reduces sore throat. H4: Gargling with green tea after surgery reduces hoarseness. H5: Impregnation of postoperative ice particles reduces hoarseness. H6: Postoperative mouthwash with arnico montana reduces hoarseness.

Research Question

1. Do ice particles impregnation, gargling with green tea and gargling with arnico montana reduce intubation-related sore throat in patients undergoing general anesthesia?
2. Do ice particles impregnation, gargling with green tea and gargling with arnico montana reduce hoarseness due to intubation in patients undergoing general anesthesia?

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the research,
* To be 18 years or older,
* To know how to read and write,
* No hearing problem,
* Not having difficulty in understanding,
* To live before the operation,
* Having experience before surgery,
* The duration of the operation is 30 minutes or more,7
* No nasogastric catheter

Exclusion Criteria:

* Having a sore throat before surgery,
* Having hoarseness before surgery,
* To have oral and neck surgery,
* Having a history of allergy,
* Having a nasogastric catheter,
* The duration of the operation is less than 30 minutes,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Stout's hoarseness evaluation form | one day
  Stout's hoarseness evaluation form maximum 0= sound normal
  minimum of 3 = complete silence, speech
visual analog scale | one day
  the visual analog scale criterion was used to evaluate sore throat. minimum 0 = no pain
  maximum 10 = severe pain

CONTACTS AND LOCATIONS:
Overall Officials: gülcan dürüst sakallı, lecturer, Principal Investigator — doğu akdeniz üniversitesi
Locations (1):
- Eastern Mediterranean University, Nursing Department, Faculty of Health Sciences, Famagusta, North Cyprus Via Mersin 10, Turkey, Ammochostos, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jafari H, Ariaeifar MR, Yazdani Charati J, Soleimani A, Nasiri Formi E. The Effect of Green Tea Gargle Solution on Sore Throat After Coronary Artery Bypass Grafting: A Randomized Clinical Trial. Anesth Pain Med. 2016 May 9;6(3):e32108. doi: 10.5812/aapm.32108. eCollection 2016 Jun. PMID 27642569
- [Background] Tsintzas D, Vithoulkas G. Treatment of Postoperative Sore Throat With the Aid of the Homeopathic Remedy Arnica montana: A Report of Two Cases. J Evid Based Complementary Altern Med. 2017 Oct;22(4):926-928. doi: 10.1177/2156587217735986. Epub 2017 Nov 2. PMID 29228804
- [Background] Bulut H, Erden S, Demir SG, Cakar B, Erdogan Z, Demir N, Ay A, Aydin E. The Effect of Cold Vapor Applied for Sore Throat in the Early Postoperative Period. J Perianesth Nurs. 2016 Aug;31(4):291-7. doi: 10.1016/j.jopan.2014.10.005. Epub 2016 Feb 24. PMID 27444760